CLINICAL TRIAL: NCT03748108
Title: A Randomized Clinical Trial Estimating the Efficacy of Bolus Administration of Intravenous Lidocaine at the Time of Abdominal Hysterectomy to Decrease Postoperative Pain
Brief Title: Bolus Administration of Intravenous Lidocaine at the Time of Abdominal Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University Hospital (Other)
Responsible Party: Principal Investigator, hany farouk, Principal Investigator, Aswan University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: aswu/275/18
Record Dates: First submitted 2018-11-18; First posted 2018-11-20 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-08

CONDITIONS: Abdominal Hysterectomy
Keywords: lidocaine; Postoperative Pain; hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

STUDY DESIGN:
Intervention Model Description: This study will be a single-center, randomized double-blind, placebo-controlled, parallel group trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participating patients, surgeons, anesthesiologists and medical investigators who will be involved in the data collection will be all blinded to the patient's group assignment until the collection of data for all cases will be complete.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lidocaine (Experimental): A bolus intravenous dose of 1.5 mg/kg lidocaine 2% over 15 s just before the induction of general anesthesia.
  Interventions: Drug: lidocaine
- Placebo (Placebo Comparator): A bolus intravenous dose of a saline placebo over 15 s just before the induction of general anesthesia.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine — a bolus intravenous dose of 1.5 mg/kg lidocaine 2% over 15 s just before the induction of general anesthesia.
  Other Names: Experimental
  Arms: lidocaine
Drug: Placebo — a bolus intravenous dose of 1.5 mg/ kg a saline placebo over 15 s just before the induction of general anesthesia.
  Other Names: Placebo Comparator
  Arms: Placebo

SUMMARY:
The objective of the study to evaluate whether a bolus administration of intravenous lidocaine decreases postoperative pain and represents an opioid-minimizing strategy after abdominal hysterectomy compared with placebo.

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is the most common gynecological operation worldwide. Some studies noticed about abused of opioids in postoperative care, led to a more adverse effect of opioids, slow recovery, prolong the length of hospitalized stay and consequently increase the unnecessary cost of treatment.

Guidelines have considered using preoperative analgesics for reducing post-operative opioids consumption, including lidocaine infusion. With its anti-inflammatory, anti-hyperalgesia and analgesic properties, intravenous perioperative lidocaine infusion (IVLI) has been used for optimal postoperative care in different surgeries and in various procedures involving hysterectomy.

Therefore, the aim of this study is to assess the efficacy of bolus administration of intravenous lidocaine at the time of abdominal hysterectomy to decrease postoperative pain and reducing morphine requirements, after TAH.

ELIGIBILITY:
Inclusion Criteria:

* Women ranging age between 35-60 years a who undergoing elective total abdominal hysterectomy

Exclusion Criteria:

* Participants had known sensitivity to lidocaine
* Participants had difficulty in intubation
* Participants were on chronic pain medication or already on long-term opioids
* Participants smokers
* Participants with disabilities who were unable to communicate pain levels
* refuse to consent

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — women undergoing abdominal hysterectomy
Enrollment: 120 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Visual analog score during movement | 30 minutes postoperative
  movement-evoked pain measurements ranging from 0 to 10, where 0 no pain and 10 maximum pain

SECONDARY OUTCOMES:
Visual analog score during rest | 24 hours post operative
  ranging from 0 to 10, where 0 no pain and 10
number of patients need Fentanyl consumption | 24 hours post operative
  number of patients need Fentanyl consumption
number of days patients stay in hospital | 4 weeks
  calculation of number of days patients stay in hospital

CONTACTS AND LOCATIONS:
Overall Officials: hany f sallam, md, Principal Investigator — Aswan University Hospital
Locations (1):
- Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided